CLINICAL TRIAL: NCT03877627
Title: The Clinical Significance of Sentinel Lymph Node Imaging Combined With Imaging Examination in Pelvic and Peritoneal Lymphadenectomy for Endometrial Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAHoWMU-CR2019-07-102
Record Dates: First submitted 2019-03-10; First posted 2019-03-15 (Actual); Last update posted 2020-10-29 (Actual); Status verified 2020-10

CONDITIONS: Endometrial Carcinoma; Lymphadenectomy
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Intervention Model Description: 60 patients who were assessed negative by sentinel lymph node imaging combined with imaging were randomized to undergo pelvic and peritoneal lymphadenectomy.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Negative 1 (No Intervention): Patients in this arm will not undergo Pelvic and Peritoneal Lymphadenectomy.
- Negative 2 (Experimental): Patients in this arm will undergo Pelvic and Peritoneal Lymphadenectomy.
  Interventions: Procedure: Pelvic and Peritoneal Lymphadenectomy

INTERVENTIONS:
Procedure: Pelvic and Peritoneal Lymphadenectomy — Patients in arm 2 will be randomized to undergo pelvic and peritoneal lymphadenectomy to treat their endometrial carcinoma.
  Arms: Negative 2

SUMMARY:
The aim of this prospective cohort study is to explore the clinical significance of sentinel lymph node imaging combined imaging examination evaluation in pelvic and peritoneal lymphadenectomy for endometrial carcinoma management.

DETAILED DESCRIPTION:
The clinical data including surgical procedure, the situation of sentinel lymph node imaging and pathological results of patients with endometrial carcinoma treated in our hospitals between April 2019 and April 2021 will be analyzed in this study to clarify the homogeneity of imaging evaluation, sentinel lymph node development evaluation and pathological results.

ELIGIBILITY:
Inclusion Criteria:

1. Females who are diagnosed with endometrial carcinoma;
2. Patients who are willing to receive primary non-reserved fertility function surgery to treat their disease;
3. Patients who are agreed to participated in this prospective cohort study.

Exclusion Criteria:

1. Patients who still have the will to have pregnancy;
2. Patients who have other diseases or heavy injuries that will interfere with the results;
3. Simultaneous participation in another clinical study with investigational medicinal product(s) or researcher thinks the subjects are not suitable for this trial.

Ages: 10 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2023-03-15 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
the number (s) of pelvic and abdominal lymph node metastasis | 1 year during the perioperative period
  the specific number of pelvic and abdominal lymph nodes that are invaded by metastatic endometrial carcinoma
the percentage (%) of pelvic and abdominal lymph node metastasis | 1 year during the perioperative period
  the specific percentage of pelvic and abdominal lymph nodes that are invaded by metastatic endometrial carcinoma
the coincidence rate (%) of pelvic and abdominal lymph node imaging, sentinel lymph node imaging and pathological diagnosis | 1 year during the perioperative period
  by performing chi-square test by SPSS 17.0，we plan to calculate the coincidence rate of three clinical examination
the effect of pelvic lymphadenectomy on the prognosis of endometrial carcinoma patients | 1 year during the perioperative period
  by setting up the control group and experimental group and conducting follow-up，we are determined to know whether pelvic lymphadenectomy would influence the prognosis of endometrial carcinoma

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-01): https://cdn.clinicaltrials.gov/large-docs/27/NCT03877627/Prot_SAP_000.pdf